CLINICAL TRIAL: NCT03777878
Title: Carbetocin Versus Oxytocin Infusion Plus Tranexamic Acid for Prevention of Postpartum Hemorrhage at Cesarean Section: A Double-Blind Randomized Clinical Trial
Brief Title: Carbetocin Versus Oxytocin Infusion Plus Tranexamic Acid During Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/186/18
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; oxytocin; carbetocin
MeSH Terms: interventions — carbetocin; Oxytocin

STUDY DESIGN:
Intervention Model Description: A Double-Blind Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Double-Blind Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbetocin plus placebo to TA and placebo to oxytocin (Active Comparator): 100 μg carbetocin ampoule or separate placebo ampoule was diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby plus two placebo ampoules to oxytocin in 500 mL of intravenous solution infusion over 15 min after delivery of the baby plus 2 placebo ampoules to TA in 100 ml saline by slow infusion
  Interventions: Drug: Carbetocin; Drug: placebo to TA; Drug: placebo to oxytocin
- oxytocin plus TA (Active Comparator): 20 IU oxytocin in 500 mL of intravenous solution infusion over 15 min after delivery of the baby plus 1gm TA in 100ml saline by slow infusion plus placebo ampoule to carbetocin will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Interventions: Drug: oxytocin; Drug: TA; Drug: placebo to carbetocin
- oxytocin plus placebo to TA and placebo to carbetocin (Active Comparator): 20 IU oxytocin in 500 mL of intravenous solution infusion over 15 min after delivery of the baby plus 2 placebo ampoules to TA in 100 ml saline by slow infusion plus placebo ampoule to carbetocin will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Interventions: Drug: oxytocin; Drug: placebo to carbetocin; Drug: placebo to TA

INTERVENTIONS:
Drug: Carbetocin — 100 μg carbetocin ampoule will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Other Names: Active Comparator
  Arms: Carbetocin plus placebo to TA and placebo to oxytocin
Drug: oxytocin — 20 IU oxytocin in 500 mL of intravenous solution infusion over 15 min after delivery of the baby
  Other Names: Active Comparator
  Arms: oxytocin plus TA; oxytocin plus placebo to TA and placebo to carbetocin
Drug: TA — 2 ampoules of TA in 100 ml saline by slow infusion
  Other Names: active comparator
  Arms: oxytocin plus TA
Drug: placebo to carbetocin — placebo ampoule to carbetocin will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Other Names: placebo comparator
  Arms: oxytocin plus TA; oxytocin plus placebo to TA and placebo to carbetocin
Drug: placebo to TA — 2 placebo ampoules to TA in 100 ml saline by slow infusion
  Other Names: placebo comparator
  Arms: Carbetocin plus placebo to TA and placebo to oxytocin; oxytocin plus placebo to TA and placebo to carbetocin
Drug: placebo to oxytocin — two placebo ampoules to oxytocin in 500 mL of intravenous solution infusion over 15 min after delivery of the baby
  Other Names: placebo comparator
  Arms: Carbetocin plus placebo to TA and placebo to oxytocin

SUMMARY:
Purpose to evaluates the effects of oxytocin infusion with or without intravenous tranexamic acid (TA) in comparison with Carbetocin for prevention of postpartum hemorrhage at a cesarean section with one or more risk factor for postpartum hemorrhage.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is potentially life-threatening and is a significant contributor to maternal mortality and morbidity especially in developing countries. The risk of PPH is much higher for women undergoing cesarean delivery (CD). Oxytocin is regarded as the gold standard uterotonic agent but only has a half-life of 4-10 min; therefore, at cesarean section oxytocin must be administered as a continuous intravenous infusion to attain sustained uterotonic activity throughout the surgical procedure and immediate postpartum period. Carbetocin is a long-acting synthetic analog of oxytocin that can be administered as a single-dose injection; intravenously administered carbetocin has a half-life of approximately 40 min.

A single intravenous bolus of carbetocin produces a tetanic uterine contraction within 2 min and persists for an average of 60 min following injection.

The aim of this study is to compare the effectiveness of combined tranexamic acid (TA) and oxytocin infusion with intravenous carbetocin for prevention of PPH in patients with risk factors during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergo elective cesarean section with one or more risk factors for PPH were the candidates for participation
* With fetal macrosomia, polyhydramnios, low insertion of the placenta, multiple gestations, prolonged labor, chorioamnionitis, past history of PPH, diabetes and high parity (5 previous deliveries).

Exclusion Criteria:

* suspected coagulopathy,
* history of coronary artery disease or hypertension,
* women with a history of hypersensitivity to carbetocin, TA or oxytocin
* general anesthesia, and
* PPH due to causes other than uterine atony.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who undergo elective cesarean section with one or more risk factors for PPH were the candidates for participation
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
The number of the patient need of additional pharmacological uterotonic. | 24 hours post operative
  calculate the number of the patient need of additional pharmacological uterotonic.

SECONDARY OUTCOMES:
estimation of intraoperative blood loss (ml) | during the operation
  measure Intraoperative blood loss in ml by gravimetric methods
amount of postoperative blood loss | 24 hours post operative
  measure amount of blood loss post operative in ml by gravimetric methods
number of patient with postpartum hemorrhage | 24 hours post operative
  calculation of the number of the patients with blood loss >1000 ml

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University, Aswān, Egypt